CLINICAL TRIAL: NCT02953392
Title: Evaluation of Implant-Abutment Interface Design on Bone and Soft Tissue Levels Around Implants Placed Using Two Different Transcrestal Sinus Floor Elevation Approaches: A Multi-Center, Double Blind, Randomized Trial
Brief Title: Implant-Abutment Interface Design on Bone and Soft Tissue Levels Around Implants Placed Using Different Transcrestal Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU College of Dentistry (Other)
Responsible Party: Principal Investigator, Ismael Khouly, Associate Director of Periodontology & Implant Dentistry, NYU College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01349
Record Dates: First submitted 2016-09-26; First posted 2016-11-02 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): Transcrestal Sinus Floor Elevation using platform switched implant with bone graft material.
  Interventions: Device: Anorganic Bovine Bone Graft Material; Device: Shelta Platform Switching Premium Implants
- Arm 2 (Active Comparator): Transcrestal Sinus Floor Elevation using platform switched implant with no bone graft material.
  Interventions: Device: Collagen Membrane; Device: Shelta Platform Switching Premium Implants
- Arm 3 (Active Comparator): Transcrestal Sinus Floor Elevation using platform matching implant with bone graft material.
  Interventions: Device: Anorganic Bovine Bone Graft Material; Device: Shelta Platform Matching Premium Implants
- Arm 4 (Active Comparator): Transcrestal Sinus Floor Elevation using platform matching implant with no bone graft material.
  Interventions: Device: Collagen Membrane; Device: Shelta Platform Matching Premium Implants

INTERVENTIONS:
Device: Anorganic Bovine Bone Graft Material — Anorganic bovine bone graft material is intended for augmentation or reconstructive treatment of the alveolar ridge, filling periodontal defects, filling defects after root resection, apicoectomy, and cystectomy, filling extraction sockets to enhance preservation of the alveolar ridge, and elevation of maxillary sinus floor.
  Arms: Arm 1; Arm 3
Device: Collagen Membrane — Collagen dental wound dressing is intended for the management of oral wounds and sores, including; dental sores, oral ulcers, periodontal surgical wounds, suture sites, burns, extraction sites, surgical wounds, and traumatic wounds.
  Arms: Arm 2; Arm 4
Device: Shelta Platform Switching Premium Implants — Shelta implant systems are intended for immediate placement and function on single tooth and/or multiple tooth applications when good primary stability is achieved, with appropriate occlusal loading, in order to restore chewing function.
  Arms: Arm 1; Arm 2
Device: Shelta Platform Matching Premium Implants — Shelta implant systems are intended for immediate placement and function on single tooth and /or multiple tooth applications when good primary stability is achieved, with appropriate occlusal loading, in order to restore chewing function.
  Arms: Arm 3; Arm 4

SUMMARY:
Sixty patients with partially edentulous posterior maxilla requiring a transcrestal sinus floor elevation technique to insert one implant will be selected. The purpose of this multi-center, prospective, double blind, and randomized investigation is to analyze a platform switched implant when placed at limited maxillary residual bone height with low bone density compared to a platform matching implant with or without bone graft material.

DETAILED DESCRIPTION:
Approximately 60 subjects who require at least one posterior maxilla implant in the areas of the second pre-molars or (first or second) molars with 6 to 9 mm of crestal bone below the sinus floor, as determined on the computerized axial tomographic (CT) scan, will be recruited for the study. Subjects will receive dental implants to replace a missing tooth (second pre-molar or first/second molar) on one side of the maxillary arch. Each subject will receive one type of implant: platform switched (PS) or platform matching (PM). Each site will receive either a bone graft material composed of anorganic bovine bone mineralized (ABBM, Bio-Oss, Geistlich Pharma) or no graft material (collagen membrane used for wound healing (Collatape, Zimmer)). At implant placement surgery and post-surgical follow-ups, the treated site will be examined, clinically measured, and radiographs and photographs will be taken.

The central hypothesis is that the mean crestal bone level for the platform switched (test implants) implants will be superior to the mean crestal bone level for the platform matching (control implants) implants when placed in limited maxillary residual bone in the posterior regions, regardless of the use of bone graft material or collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have read, understood and signed an informed consent form.
2. Subjects must be 18 to 70 years of age.
3. Subjects must be able and willing to follow study procedures and instructions.
4. Subject must maintain good oral hygiene.
5. Subjects must have a single tooth missing in the pre-molar or molar region of the maxilla (ADA tooth positions 2-4 and 13-15; FDI tooth positions 15-17 and 25-27).
6. The mesio-distal distance of the tooth gap at bone level must be at least 6.8 mm to allow for placement of the Ø3.8 mm implant with a minimal distance of 1.5 mm from the implant shoulder to the adjacent tooth at bone level. A minimum of 7.8 mm of buccal-lingual ridge to allow 2 mm of buccal and lingual plate will be required.
7. No apical disorder/inflammation at the area of the implant site.
8. Residual bone height ranging from 6 to 9 mm.
9. The implant must penetrate at least 2 mm into the sinus on the mesial or distal sides.
10. Sufficient bone width in the edentulous region (≥ 6mm).
11. Subjects must be committed to the study and attend the required follow-up visits.

Exclusion Criteria:

1. Subjects with a systemic disease that would preclude dental implant surgery (e.g. serious internal medical problems, disorders of bone metabolism, uncontrolled bleeding disorders, weakened immune system, illness requiring periodic use of steroids, uncontrollable endocrine disorders, uncontrolled diabetes).
2. Subjects who have failed to maintain good plaque control.
3. Subjects with any contraindications for oral surgical procedures (e.g. inadequate wound healing capacity, poor oral hygiene, maxillary and mandibular growth not completed, xerostomia).
4. Subjects with mucosal diseases (e.g., erosive lichen planus) in the localized area around the study implant site.
5. Subjects presenting with maxillary sinus pathology.
6. Subjects with a history of local irradiation therapy in the head/neck region.
7. Subjects with severe bruxing, parafunctional habits, or temporomandibular joint dysfunction.
8. Subjects receiving, or having a history of receiving intravenous or subcutaneous antiresorptive agents associated with osteonecrosis of the jaw, such as bisphosphonates.
9. Oblique sinus floor (> 45 inclination).
10. Subjects with any untreated endodontic lesions or untreated periodontal disease.
11. Subjects who are heavy smokers (defined as >10 cigarettes per day or >1 cigar per day) or chew tobacco, including within 3 months prior to enrollment.
12. Subjects who have physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene.
13. Subjects who are pregnant or intending to become pregnant during the duration of the study.
14. Subjects requiring bone augmentation or socket grafting prior to surgery.
15. Subject allergic to collagen or porcine derived products.
16. Subjects with conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non- compliance or unreliability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Mean crestal bone level changes measured in mm using periapical radiographs and CT scans. | 12 months
  Mean crestal bone level change around the implants will be determined by periapical radiographs of mesial and distal bone levels. CT scans will be used to determine buccal and lingual bone level change between implant placement and 12 months, following placement of a platform switched implants or platform matching implants.
Mean periapical sinus bone level changes measured in mm using periapical radiographs and CT scans. | 12 months
  Mean periapical sinus bone level change between implant placement and 12 months will be determined by radiographic measurement (using periapical radiographs and CT scans) following placement of a platform switched implant or platform matching implant in the posterior region of the maxilla, with bone graft material or without bone graft material.
Implant survival measured through observation. | 12 months
  Implant survival will be measured at implant loading and 12 months following implant placement will be assessed through clinical observation.
Implant success rate measured by percentage. | 12 months
  Implant success rate will be assessed at implant loading and 12 months following implant placement measured by percentage.

SECONDARY OUTCOMES:
Crestal bone height changes measured in mm using periapical radiographs. | 12 months
  Additional crestal bone height change determined by measurements of periapical radiographs of mesial and distal bone levels between implant placement and implant loading, and between implant loading and 12 months post-implant placement.
Implant Stability Quotient (ISQ) measured in N/cm. | 6 months
  Implant Stability Quotient (ISQ) between implant placement and implant loading and at 6 months and between implant loading.
Periodontal Pocket Depths measured in mm. | 12 months
  Periodontal Pocket Depths assessed at screening, implant loading, and 12 months post-implant placement.
Subject satisfaction assessed through questionnaire. | 12 months
  Subject satisfaction at implant placement, immediate post-operative, and 12 months post-implant placement.
Changes in sinus anatomy measured in mm compared to implant survival. | 12 months
  Changes in the sinus anatomy measured in mm compared to implant survival.
Changes in sinus anatomy measured in mm compared to implant success. | 12 months
  Changes in the sinus anatomy measured in mm compared to implant success.
Changes in sinus anatomy measured in mm compared to crestal bone changes. | 12 months
  Changes in the sinus anatomy measured in mm compared to crestal bone level changes. implant stability (ISQ).
Changes in sinus anatomy measured in mm compared to implant stability. | 12 months
  Changes in the sinus anatomy measured in mm compared to implant stability (ISQ).
Changes residual crestal bone height measured in mm compared to implant survival. | 12 months
  Changes in residual crestal bone height compared to implant survival.
Changes residual crestal bone height measured in mm compared to implant success. | 12 months
  Changes in residual crestal bone height compared to implant success.
Changes residual crestal bone height measured in mm compared to implant stability. | 12 months
  Changes in residual crestal bone height compared to implant stability (ISQ).
Changes residual crestal bone height measured in mm compaierd to sinus bone levels. | 12 months
  Changes in residual crestal bone height compared to sinus bone levels.
Bleeding on probing measured by present or not present. | 12 months
  Bleeding on probing assessed at screening, implant loading, and 12 months post-implant placement.
Gingival Recession measured in mm. | 12 months
  Gingival recession assessed at screening, implant loading, and 12 months post-implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael E Khouly, DDS, MS, PhD, Principal Investigator — Bluestone Center for Clinical Research
Locations (1):
- Bluestone Center for Clinical Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No